CLINICAL TRIAL: NCT04212273
Title: A Single-center, Prospective Controlled Study of the Diagnostic Efficacies of Sonazoid-CEUS and EOB-MRI in Patients With High Risk of HCC
Brief Title: Diagnostic Efficacies of Sonazoid-CEUS and EOB-MRI in Patients With High Risk of HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Third Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: drjingxiang001
Record Dates: First submitted 2019-12-02; First posted 2019-12-26 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Cancer; Liver Cirrhoses; Diagnoses Disease
Keywords: Hepatocellular carcinoma; Sonazoid Contrast-enhanced ultrasound; EOB-MRI; Diagnostic Efficacy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Sonazoid-CEUS and EOB-MRI (Experimental): Patients with high risk of HCC having suspicious lesions on US will receive Sonazoid-CEUS and EOB-MRI examinations.
  Interventions: Diagnostic Test: Diagnostic Sonazoid-CEUS and EOB-MRI

INTERVENTIONS:
Diagnostic Test: Diagnostic Sonazoid-CEUS and EOB-MRI — Undergo Sonazoid-CEUS and EOB-MRI

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer. Patients with HCCs usually have a poor prognosis. Hepatocarcinogenesis is an intricate and multistep process. Detecting and staging early HCC in patients with liver cirrhosis are still challenging for imaging techniques. Contrast-enhanced ultrasonography (CEUS) and gadoxetic acid-enhanced magnetic resonance imaging (EOB-MRI) are widely used in clinical practice. EOB-MRI has advantages of high detecting rate for small lesions, high sensitivity of hepatobiliary phase and extensive image information. Sonazoid has the advantage of offering a unique post-vascular phase, also called the Kupffer phase. Therefore, malignant tumors with few or no Kupffer cells appear as contrast defects, with respect to the relatively well-enhanced surrounding liver in the postvascular phase. The diagnostic efficacies of these two imaging methods have not been well studied. Therefore, the purpose of this study is to compare the efficacies of Sonazoid-CEUS and EOB-MRI in patients with high risk of HCC, and to compare the detection ability for malignant tumors by Kupffer phase and hepatobiliary phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are at high risk for HCC.
2. The ages of patients are between 18 and 80.
3. Patients are with solid liver lesion(s) detected by US: if a patient has a solitary tumor, the size of the tumor is less than or equal to 5 cm; if a patient has multiple lesions, the sizes of the tumors are less than or equal to 3 cm and the number of lesions is less than or equal to 3.
4. Patient is able and willing to receive CEUS and EOB-MRI examinations within 30 days.
5. Patient signs the informed consent. -

Exclusion Criteria:

1. Patient is with lesions confirmed by pathology or follow-up, or hemangiomas.
2. Patient is with lesions already undergoing local treatment, including thermal ablation or TACE.
3. Patient is with severe cardiopulmonary insufficiency.
4. Patient is a pregnant or breastfeeding women.
5. Patient is considered to be unsuitable to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-21 (Actual); Primary Completion 2022-12-24 (Estimated); Study Completion 2022-12-24 (Estimated)

PRIMARY OUTCOMES:
The sensitivity, specificity and accuracy of Sonazoid-CEUS and EOB-MRI | 6 to 12 months
  The sensitivity, specificity and accuracy of Sonazoid-CEUS and EOB-MRI in the diagnosis for patients with high risk of HCC will be determined.

SECONDARY OUTCOMES:
The detection rate of the additionally found HCC | 6 to 12 months
  The detection rate of the additionally found HCC on Sonazoid-CEUS and EOB-MRI will be determined .

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Jing, MD, Study Director — Tianjin Third Central Hospital
Locations (1):
- Tianjin Third Central Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for the Study of the Liver. Corrigendum to "EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma" [J Hepatol 69 (2018) 182-236]. J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. Epub 2019 Feb 7. No abstract available. PMID 30739718
- [Background] Omata M, Cheng AL, Kokudo N, Kudo M, Lee JM, Jia J, Tateishi R, Han KH, Chawla YK, Shiina S, Jafri W, Payawal DA, Ohki T, Ogasawara S, Chen PJ, Lesmana CRA, Lesmana LA, Gani RA, Obi S, Dokmeci AK, Sarin SK. Asia-Pacific clinical practice guidelines on the management of hepatocellular carcinoma: a 2017 update. Hepatol Int. 2017 Jul;11(4):317-370. doi: 10.1007/s12072-017-9799-9. Epub 2017 Jun 15. PMID 28620797
- See also: HCC diagnosis guideline — https://linkinghub.elsevier.com/retrieve/pii/S0168-8278(19)30034-0
- See also: HCC diagnosis guideline — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5491694/
- See also: EOB-MRI — https://link.springer.com/article/10.1007/s00330-010-2030-1